CLINICAL TRIAL: NCT02824003
Title: Double Blind, Randomized, Placebo-Controlled, Phase 2A Mechanistic Study to Evaluate the Effect of ISIS 449884 (ISIS-GCGRRx) on Hepatic Lipid and Glycogen Content in Patients With Type 2 Diabetes Being Treated With Metformin
Brief Title: Study to Evaluate the Effect of ISIS GCGRRx on Hepatic Lipid and Glycogen Content in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 449884-CS3
Record Dates: First submitted 2016-06-15; First posted 2016-07-06 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISIS-GCGRRx (Experimental): ISIS-GCGRRx once weekly dosing for 13 weeks
  Interventions: Drug: ISIS-GCGRRx
- Placebo (Placebo Comparator): once weekly dosing for 13 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISIS-GCGRRx — once weekly dosing for 13 weeks
  Other Names: ISIS 449884
  Arms: ISIS-GCGRRx
Drug: Placebo — once weekly dosing for 13 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of ISIS 449884 (ISIS-GCGRRX) on Hepatic Lipid and Glycogen Content in patients with Type 2 Diabetes being treated with Metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 75
* BMI ≥ 25.0 kg/m2 < 36.0 kg/m2
* HbA1c ≥ 7.5% and ≤ 10.5%
* Type 2 Diabetes Mellitus and on stable dose of Metformin. Patients must have been on a stable dose of oral metformin (at least 1000 mg/day) for a minimum of 3 months prior to screening evaluation and will be required to continue their stable dose of metformin throughout the study. Patients on a stable dose of metformin plus a sulfonylurea (SU) or metformin plus a dipeptidyl peptidase-IV (DPPIV) inhibitor for a minimum of 3 months prior to Screening evaluation may be allowed
* Agree to conduct home-based (fasted) blood glucose testing as directed

Exclusion Criteria:

* Clinically significant abnormalities in medical history or physical exam
* Show evidence of uncorrected hypothyroidism or hyperthyroidism
* History of liver transplantation or renal dialysis
* History of liver disease
* History of greater than 3 episodes of severe hypoglycemia within 6 months of screening
* Treatment with any other antidiabetic drug(s) other than metformin, SU or DPPIV within 3 months of screening
* History of diabetic ketoacidosis
* Any other significant illness or condition that may interfere with the patient participating or completing the study
* Inability or unwillingness to comply with protocol or study procedures -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Change in fasting hepatic glycogen content | Week 14
  Change from Baseline
Change in fasting hepatic lipid content | Week 14
  Change from Baseline

SECONDARY OUTCOMES:
Safety and Tolerability will be assessed by determining the incidence, severity, dose relationship of adverse effects, and changes in laboratory evaluations | 38 weeks
  Safety results in patients dosed with ISIS 449884 will be compared with those from patients dosed with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Bhanot, Study Director — Ionis Pharmaceuticals
Locations (1):
- Ionis Investigator Site, Vienna, Austria

REFERENCES:
- [Derived] Morgan ES, Tai LJ, Pham NC, Overman JK, Watts LM, Smith A, Jung SW, Gajdosik M, Krssak M, Krebs M, Geary RS, Baker BF, Bhanot S. Antisense Inhibition of Glucagon Receptor by IONIS-GCGRRx Improves Type 2 Diabetes Without Increase in Hepatic Glycogen Content in Patients With Type 2 Diabetes on Stable Metformin Therapy. Diabetes Care. 2019 Apr;42(4):585-593. doi: 10.2337/dc18-1343. Epub 2019 Feb 14. PMID 30765435